CLINICAL TRIAL: NCT03339505
Title: Salovum (Antisecretory Factor) in Patients With Severe Traumatic Brain Injury
Brief Title: Effect of Antisecretory Factor, Given as a Food Supplement to Adult Patients With Severe Traumatic Brain Injury
Acronym: SASAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peter Siesjö (Other)
Collaborators: University of Stellenbosch (Other)
Responsible Party: Sponsor-Investigator, Peter Siesjö, Professor, Consultant, Skane University Hospital
Organization: Skane University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ethics Reference #: M16/10/040
Record Dates: First submitted 2017-09-20; First posted 2017-11-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Brain Trauma
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded and prospective.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded until the end of the trial. Unmasking will take place once all patients are included and the trial is concluded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): Patients in treatment group will receive Salovum according to g/kg body weight/24 hours/divided into 6 doses, during a maximum of 5 days
  Interventions: Dietary Supplement: Salovum
- Placebo group (Placebo Comparator): Patients in treatment group will receive Placebo (egg yolk powder) according to g/kg body weight/24 hours/divided into 6 doses, during a maximum of 5 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Salovum — Dietary supplement with high concentration of anti-secretory factor
  Arms: Treatment group
Dietary Supplement: Placebo — Placebo for Salovum
  Arms: Placebo group

SUMMARY:
The present trial intends to assess whether Salovum®, an egg powder enriched for antisecretory factor given to patients with severe traumatic brain injury will improve outcome compared to a control group given placebo egg powder.

100 patients with GCS<9 will be enrolled and randomised to active or placebo treatment during maximum 5 days. Salovum® or placebo will be administered orally by nasogastric feeding tubes.

Primary endpoint will be overall 30 data mortality. Secondary endpoints will be intracranial pressure and treatment intensity level.

DETAILED DESCRIPTION:
Treatment of increased ICP, using Anti-secretory Factor, in patients with severe head trauma Brain edema, defined as an increased fluid content in either the extracellular or intracellular space, arise in both trauma and in conjunction with other brain pathologies such as infectious diseases, intracranial tumors and ischemic events, i.e. stroke. The mechanisms underlying the formation of edema are not fully understood. In the injured brain, leakage over the blood brain-barrier arise which leads to transport of fluid from the blood to the extracellular space, causing an extracellular or vasogenic edema. Damage to cell membranes and disruption of cell function causes an intracellular or cytotoxic edema. Although one type of edema may predominate initially, one type most likely leads to another. In addition to the physiological, flow-related changes that arise, the edema is also worsened by the inflammatory response to damage. In the injured brain, disease associated molecular patterns (DAMP), and pro-inflammatory cytokines that can give rise to both intracellular and extracellular edema are released.

If the edema becomes expansive enough to give rise to a significant increase in intracranial pressure the circulation of the brain is threatened and surgical intervention inevitable. The most common procedure is hemicraniectomy, a procedure intended to add more space for the edematous brain to expand. The procedure itself is risky, and re-operations due to hematoma, CSF-leakage and more are common. Furthermore, it is not known how the procedure itself affects the brain in terms of increased edema, tearing of the brain etc.

Antisecretory factor, AF is a 41 kDa protein that exists in most mammals. It was first discovered due to its ability to inhibit experimental diarrhea. Endogenous AF secretion increases after exposure to bacterial toxins and an increase in AF secretion in combination with an inflammatory reaction may be a part of normal defense against the secretory and inflammatory component in diarrhea and other pathological processes involving membrane leakage and inflammation. AF has been shown to modulate pro-inflammatory and anti- inflammatory cytokine release. AF has also been shown to be effective against vertigo symptoms in Meniere's disease, which is believed to be caused by an abnormal collection of lymph around the balance nerve. AF and AF16 (the functional terminal 16 amino-acid peptide) have been tested in animal models of cerebral edema such as herpes encephalitis and traumatic brain injury with significant reduction of intracranial pressure, morbidity and mortality AF is commercially available for human use as Salovum®, an egg yolk powder B221® enriched for AF. It is available in pharmacies without prescription, but can also be prescribed as a dietary supplement in Sweden. Salovum® is classified as a "medical food" by the Swedish Pharmaceutical Agency and the European Union. Salovum® is currently registered in the Republic of South Africa.

Hypothesis Cerebral edema in traumatic brain injury is caused by inflammation triggered by tissue damage. The anti-secretory and anti-inflammatory compound Salovum® has the potential to counteract this and thus reduce cerebral edema in traumatic brain injury. Furthermore, the reduction of cerebral edema is hypothesized to decrease intracranial pressure, reduce the development of secondary brain damage and subsequently reduce treatment intensity levels and death.

Aims and Objectives Though, the number of patients with severe traumatic head injury in Sweden is decreasing and the need for a larger, randomized trial in a centre with large volumes of traumatic brain injury is needed The primary focus for scientific investigation is to evaluate if AF given as a dietary supplement (Salovum®) will reduce 30-day mortality in adult patients with severe traumatic brain injury. The secondary aims are to investigate whether AF will reduce intracranial pressure and treatment intensity levels - TIL, during intervention.

Methodology The outlined study is a phase-2, prospective, double-blinded, randomized, placebo-controlled trial. After inclusion patients will be randomized to active Salovum® or placebo egg powder treatment every 4th hour during 5 days. Treatment of patients will be according to current algorithms at the study site.

Study population 100 adult (age 18+) patients with severe traumatic brain injury, where ICP-monitoring is deemed necessary, will be included in the study.

Patient samples A venous whole blood sample will be drawn before and after treatment in all patients. The blood sample will be frozen and stored at the study site for further analysis.

Anticipated benefits In an ongoing Swedish study, preliminary results indicate that AF has a very potent ICP- lowering effect in patients with severe TBI and other pathologies encompassing cerebral edema, which might prove an effect on 30-day mortality in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adult of either gender between 18 and 65 years.
2. Non-penetrating, isolated severe traumatic brain injury
3. GCS >3 and GCS<9 on admission or within 48 hours after injury*
4. Admission to study hospital within 24 hours of injury*
5. No known history of allergy to egg-protein
6. Planned for intracranial pressure monitoring
7. Absence of bilaterally dilated pupils
8. CT scan with traumatic pathology that is more than an isolated epidural hematoma

   * Within 24 hours of injury (for patients with GCS < 9 on admission) or Within 24 hours of deterioration (among patients deteriorating to GCS < 9 within 48 hours of injury)

Exclusion Criteria:

1. No consent 2. Systolic blood pressure below 90 mm Hg post resuscitation 3. Epidural hematoma with no other signs of intra-cranial injury 4. Penetrating injury 5. Non-fulfillment of inclusion criteria after screening and inclusion procedures.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-17 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
30 day mortality | 30 days
  Death within 30 days of trauma

SECONDARY OUTCOMES:
TIL - Treatment Intensity Level | 0-5 days
  TIL is scored at the end of each 24 hour period in the NICU, where 0 is lowest intensity and 38 is maximum intensity
ICP - Intracranial Pressure | 0-5 days
  ICP in mm Hg is recorded every hour during 0-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan J Vlok, Professor, Principal Investigator — University of Stellenbosch
Locations (1):
- Department of Neurosurgery, Tygerberg Hospital, Francie Van Zijl Dr, Cape Town, South Africa

REFERENCES:
- [Background] Eide PK, Eidsvaag VA, Hansson HA. Antisecretory factor (AF) exerts no effects on intracranial pressure (ICP) waves and ICP in patients with idiopathic normal pressure hydrocephalus and idiopathic intracranial hypertension. J Neurol Sci. 2014 Aug 15;343(1-2):132-7. doi: 10.1016/j.jns.2014.05.054. Epub 2014 Jun 2. PMID 24928077
- [Background] Zaman S, Aamir K, Lange S, Jennische E, Silfverdal SA, Hanson LA. Antisecretory factor effectively and safely stops childhood diarrhoea: a placebo-controlled, randomised study. Acta Paediatr. 2014 Jun;103(6):659-64. doi: 10.1111/apa.12581. Epub 2014 Mar 10. PMID 24484450
- [Background] Leong SC, Narayan S, Lesser TH. Antisecretory factor-inducing therapy improves patient-reported functional levels in Meniere's disease. Ann Otol Rhinol Laryngol. 2013 Oct;122(10):619-24. PMID 24294684
- [Background] Alam NH, Ashraf H, Olesen M, Salam MA, Gyr N, Meier R. Salovum egg yolk containing antisecretory factor as an adjunct therapy in severe cholera in adult males: a pilot study. J Health Popul Nutr. 2011 Aug;29(4):297-302. doi: 10.3329/jhpn.v29i4.8443. PMID 21957667
- [Background] Ulgheri C, Paganini B, Rossi F. Antisecretory factor as a potential health-promoting molecule in man and animals. Nutr Res Rev. 2010 Dec;23(2):300-13. doi: 10.1017/S0954422410000193. Epub 2010 Aug 5. PMID 20684797
- [Background] Hanner P, Rask-Andersen H, Lange S, Jennische E. Antisecretory factor-inducing therapy improves the clinical outcome in patients with Meniere's disease. Acta Otolaryngol. 2010 Feb;130(2):223-7. doi: 10.3109/00016480903022842. PMID 19479454
- [Background] Zaman S, Mannan J, Lange S, Lonnroth I, Hanson LA. B 221, a medical food containing antisecretory factor reduces child diarrhoea: a placebo controlled trial. Acta Paediatr. 2007 Nov;96(11):1655-9. doi: 10.1111/j.1651-2227.2007.00488.x. PMID 17937690
- [Background] Laurenius A, Wangberg B, Lange S, Jennische E, Lundgren BK, Bosaeus I. Antisecretory factor counteracts secretory diarrhoea of endocrine origin. Clin Nutr. 2003 Dec;22(6):549-52. doi: 10.1016/s0261-5614(03)00057-8. PMID 14613757
- [Background] Al-Olama M, Lange S, Lonnroth I, Gatzinsky K, Jennische E. Uptake of the antisecretory factor peptide AF-16 in rat blood and cerebrospinal fluid and effects on elevated intracranial pressure. Acta Neurochir (Wien). 2015 Jan;157(1):129-37. doi: 10.1007/s00701-014-2221-7. Epub 2014 Sep 24. PMID 25248325
- [Background] Al-Olama M, Wallgren A, Andersson B, Gatzinsky K, Hultborn R, Karlsson-Parra A, Lange S, Hansson HA, Jennische E. The peptide AF-16 decreases high interstitial fluid pressure in solid tumors. Acta Oncol. 2011 Oct;50(7):1098-104. doi: 10.3109/0284186X.2011.562240. Epub 2011 Mar 4. PMID 21375367
- [Derived] Cederberg D, Harrington BM, Vlok AJ, Siesjo P. Effect of antisecretory factor, given as a food supplement to adult patients with severe traumatic brain injury (SASAT): protocol for an exploratory randomized double blind placebo-controlled trial. Trials. 2022 Apr 23;23(1):340. doi: 10.1186/s13063-022-06275-z. PMID 35461285